CLINICAL TRIAL: NCT00880451
Title: Development and Decline of Brain and Cognition Through the Life Span
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909027; 09-M-N027
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2012-09

CONDITIONS: Alzheimer's Disease
Keywords: Children and Adolescents; Aging; Brain Imaging; MRI (Magnetic Resonance Imaging); MRI; Magnetic Resonance Imaging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The protocol objectives are to enable prospective IRB review of research using human MRI scans and data collected under other branch protocols or extramural sources. By combining data from multiple sources the investigators will be able to conduct analyses that require large numbers of observations that exceed the numbers collected in any single study. They will also be able to stratify and subgroup the combined samples in different ways to permit analyses that would otherwise not be possible. The study population consists of normal individuals and clinical groups of all ages. Clinical groups will be added by amendment including patients suffering from schizophrenia, ADHD, autism, Klinefelter's disease, and Alzheimer's disease. The study design consists of 1) automated segmentation of MRI brain scans to obtain regional measurements of cortical thickness and volumetric measurements of brain structures including basal ganglia, 2) manual segmentation of brain structures and brain anomalies not amenable to automated segmentation such as Virchow-Robbins spaces, 3) correlation analyses between MRI brain measurements and available demographic (e.g. gender) and physiological (e.g. BMI) data, statistical analysis of group differences where the groups are defined by diagnosis, age, gender or by other potentially useful classification. Since all data were collected under other protocols there are no additional risks or benefits associated with this protocol. This protocol combines MRI data from disparate sources and can provide important information regarding factors that may affect the comparability of MRI scans obtained from different sites using various types of MRI scanners and pulse sequences to generate MRI images. It will also enable the analysis of specific subgroups with sufficient numbers of observations for meaningful statistics.

DETAILED DESCRIPTION:
The protocol objectives are to enable prospective IRB review of research using human MRI scans and data collected under other branch protocols or extramural sources. By combining data from multiple sources, the investigators will be able to conduct analyses that require large numbers of observations that exceed the numbers collected in any single study. They will also be able to stratify and subgroup the combined samples in different ways to permit analyses that would otherwise not be possible. The study population consists of normal individuals and clinical groups of all ages. Clinical groups will be added by amendment, including patients suffering from schizophrenia, ADHD, autism, Klinefelter's disease, and Alzheimer's disease. The study design consists of 1) automated segmentation of MRI brain scans to obtain regional measurements of cortical thickness and volumetric measurements of brain structures including basal ganglia, 2) manual segmentation of brain structures and brain anomalies not amenable to automated segmentation such as Virchow-Robbins spaces, 3) correlation analyses between MRI brain measurements and available demographic (e.g. gender) and physiological (e.g. BMI) data, statistical analysis of group differences where the groups are defined by diagnosis, age, gender or by other potentially useful classification. Since all data were collected under other protocols there are no additional risks or benefits associated with this protocol. This protocol combines MRI data from disparate sources and can provide important information regarding factors that may affect the comparability of MRI scans obtained from different sites using various types of MRI scanners and pulse sequences to generate MRI images. It will also enable the analysis of specific subgroups with sufficient numbers of observations for meaningful statistics.

ELIGIBILITY:
* Data Analysis Only

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2009-03

CONTACTS AND LOCATIONS:
Overall Officials: Francois M Lalonde, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health (NIMH), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-M-0198.html